CLINICAL TRIAL: NCT04286685
Title: Development of a New Prognostic Assessment Tool for Postoperative Myocardial Injury : the TROPUTILE Score. A Non-interventional Prospective Study
Brief Title: Development of a New Prognostic Assessment Tool for Postoperative Myocardial Injury
Acronym: TROPUTILE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC19.0202 (TROPUTILE)
Record Dates: First submitted 2020-02-25; First posted 2020-02-27 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2023-12

CONDITIONS: Perioperative Complication; Myocardial Injury
Keywords: Non cardiac surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Myocardial injury after noncardiac surgery (MINS) is common, silent, and strongly associated with morbi-mortality.

There are some evidences in the littérature showing that troponin elevation pre and/or postoperatively and surgical Apgar score are strongly and independently associated with postoperative morbi-mortality.

In this cohort study of orthopedic surgery patients (> 50years), the aim is to determine MINS incidence and to assess wich peri-operative factors are associated with the occurrence of MINS. The final objective is to create a score to better identified the patients with a MINS and a poor outcome.

ELIGIBILITY:
Inclusion Criteria:

* > 50 years
* orthopedic surgery (hip, knee, spine)
* written consent

Exclusion Criteria:

* no troponin measurement prior surgery
* sepsis
* acute coronary syndrome
* pulmonary embolism
* refusing to participate
* guardianship

Ages: 50 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients aged of 50 years and more, with elective orthopedic surgery in Brest community-affiliated hospital
Sampling Method: Probability Sample
Enrollment: 1600 (Estimated)
Dates: Start 2020-01-07 (Actual); Primary Completion 2025-04-07 (Estimated); Study Completion 2025-04-07 (Estimated)

PRIMARY OUTCOMES:
Postoperative MINS incidence | 3 days after surgery
  Troponin elevation > 5ng/l compared to previous measurement OR troponin elevation > 65 ng/l

SECONDARY OUTCOMES:
Number of Participants with cardiac arrest | 3 months
  Cardiac arrest
Number of Participants with an episode of acute pulmonary oedema | 3 months
  Acute pulmonary oedema
Number of Participants with coronary angioplasty | 3 months
  Coronary angioplasty
Number of Participants with myocardial infarction | 3 months
  Myocardial infarction
Number of Participants with stroke | 3 months
  Stroke
Number of Participants with transient stroke | 3 months
  Transient stroke
Mortality rate | 3 months
  Death
Revised Cardiac Risk Index for Pre-Operative Risk (Lee score) | Inclusion
  Minimum value = 0 Minimum value = 0, maximum value = 6, higher scores mean a worse outcome (higher peri operative mortality risk)
Metabolic Equivalent of Task (MET) | Inclusion
  Minimum value = 1, Maximum value= 10, a low score (MET <4) is associated with a capacity to do some light intensity activities and is associated with cardiovascular risk.

CONTACTS AND LOCATIONS:
Overall Officials: Olivier HUET, MD, PhD, Principal Investigator — CHRU Brest
Locations (2):
- France (2):
  - CHRU Brest, Brest
  - CHU Rennes, Rennes

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning 21 months and ending five years following the publication
Access Criteria: Data access requests will be reviewed by the international committee of Brest UH . Requestors will be required to sign and complete a data acess agreement